CLINICAL TRIAL: NCT00554892
Title: ClinicalTrial in Rectal Cancer Surgery Without Mechanical Bowel Preparation
Brief Title: Rectal Cancer Surgery Without Mechanical Bowel Preparation
Acronym: PREPACOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cécile Jourdain, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060233; AOM 06086; IDRCB 2007-A00471
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Patients With Rectal Cancer
Keywords: Rectal cancer; Sphincter preservation; Mechanical bowel preparation; Post operative morbidity; Anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak | interventions — Cathartics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bowel preparation
  Interventions: Procedure: bowel preparation
- 2 (Experimental): without bowel preparation
  Interventions: Procedure: no preparation bowel

INTERVENTIONS:
Procedure: bowel preparation — oral laxatives, retrograde enemas
  Arms: 1
Procedure: no preparation bowel — no preparation bowel
  Arms: 2

SUMMARY:
The aim of this controlled multicentric study is to assess rectal cancer surgery with sphincter preservation without pre operative mechanical bowel preparation

DETAILED DESCRIPTION:
Preoperative mechanical bowel preparation (MBP) (i.e. including oral laxatives, retrograde enemas and/or oral diet before surgery) is the standard practice in colorectal surgery. The importance of MBP in preventing anastomotic leakage and infectious morbidity after elective colorectal surgery has been a dogma among surgeons for many years. The main reason is the belief that postoperative complications is related to septic bowel content. However, there is a paucity of scientific evidence demonstrating the efficacy of this practice in reducing morbidity. Moreover, potential disadvantages of MBP include the requirement for a longer preoperative duration of admission before surgery, its time consuming nature, being expensive and unpleasant for the patient and expose the early population to the particular risk of fluid and electrolyte imbalance .At least eight randomized clinical trials and two meta-analyses failed to show any superiority of MBP in colorectal surgery. On the contrary, they demonstrated that preparation might lead to an increased rate of septic complications. Such initial dates lead surgeons to re-evaluate their current clinical practice in colonic surgery. But to dates, these findings cannot finally be applied to rectal surgery because of insufficient dates. To date, no study about MBP was specifically devoted to rectal surgery. Moreover, it is currently admitted that the risk of septic complications following rectal resection, as a result of the well-known risk factors, is higher than after colonic preparation. It is the reason why most of the colorectal surgeons consider that a no preparation regimen in rectal cancer surgery could represent an additive risk factor for postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* patient with rectal cancer without any metastasesRectal excision with sphincter preservation with colorectal or coloanal anastomosis (with or without temporary ileostomy)

Exclusion Criteria:

* Stage IV disease
* Comorbidity with post operative infectious risk corticoids,immunodeficiency, Crohn's disease, ulcerative colitis ...)
* Abdominoperineal resection
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Overall morbidity including infectious and non infectious complications | peri operative

SECONDARY OUTCOMES:
- peri operative mortality - non infectious morbidity - anastomotic leakage - hospital stay - per operative evaluation of bowel preparation - clinical evaluation of bowel preparation | 30 days, 6 months
Evaluate the postoperative complications classified according to the DINDO classification. | during the study

CONTACTS AND LOCATIONS:
Overall Officials: PANIS Yves, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - CHU, Angers
  - Hopital Saint André, Bordeaux
  - Hopital Ambroise Paré, Boulognes Billancourt
  - CHU, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hopital Nord, Marseille
  - Institut Paoli Calmette, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Hopital Cochin, Paris
  - CHU Purpan, Toulouse
  - CHRU Trousseau, Tours

REFERENCES:
- [Derived] Bretagnol F, Panis Y, Rullier E, Rouanet P, Berdah S, Dousset B, Portier G, Benoist S, Chipponi J, Vicaut E; French Research Group of Rectal Cancer Surgery (GRECCAR). Rectal cancer surgery with or without bowel preparation: The French GRECCAR III multicenter single-blinded randomized trial. Ann Surg. 2010 Nov;252(5):863-8. doi: 10.1097/SLA.0b013e3181fd8ea9. PMID 21037443